CLINICAL TRIAL: NCT06267196
Title: The Effect of the Stress Ball Used During Spinal Anesthesia on Pain and Anxiety
Acronym: stressball
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Özge Sayın Ayan, Principal Investigator, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CemilTascıogluERHO-AYAN
Record Dates: First submitted 2023-12-14; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Pain; Anxiety
Keywords: Stress; Spinal anesthesia
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball group (Active Comparator): The patient group in which a stress ball is used during spinal anesthesia.
  Interventions: Other: The use of a stress ball
- The control group (No Intervention): The group that receives only standard spinal anesthesia

INTERVENTIONS:
Other: The use of a stress ball — The effect of the stress ball used during spinal anesthesia on pain and anxiety
  Arms: Stress ball group

SUMMARY:
The aim is to determine the impact of the stress ball used during spinal anesthesia on pain and anxiety levels

DETAILED DESCRIPTION:
Our planned study, which is intended to be conducted as a prospective randomized controlled trial, will include patients aged 18 and above who fall into category 3 and 4 according to the classification used in the study by Lucas et al., and who are undergoing cesarean section.Patient data including age, weight, height, body mass index (BMI), ASA (American Society of Anesthesiologists) score, gravidity, parity, history of abortion, gestational age, medical history, and surgical history will be recorded.The anxiety status of patients will be recorded using the State Anxiety Inventory (STAI-I) score both before and after the procedure.Patients will be divided into two groups using a randomization method. One group will be provided with a stress ball to squeeze during the administration of spinal anesthesia, while the second group will undergo spinal anesthesia without receiving a stress ball.All patients will receive intrathecal injection of 0.05% bupivacaine using a 25-gauge spinal needle. The Visual Analog Scale (VAS) will be assessed and recorded during the procedure to evaluate the patients' pain status.Additionally, the patient's blood pressure, pulse, and saturation levels will be recorded before starting the procedure and 2 minutes after the procedure initiation. Patient satisfaction will be evaluated after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and above.
* Patients with cesarean category 3 and 4.

Exclusion Criteria:

* Patients under the age of 18
* Patients undergoing emergency cesarean section
* Patients with bleeding disorders
* Individuals with psychological disorders

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Our study will be conducted in pregnant patients.
Enrollment: 140 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
stress ball and anxiety | Before and after the procedure, at 5 minutes.
  The impact of stress ball use during spinal anesthesia on anxiety.The effect will be assessed with the STAI (State-Trait Anxiety Inventory)scale both before and after the procedure. On this scale, the minimum and maximum values range between 20 and 80, and higher values indicate greater stress.
stress ball and pain | during the procedure
  Evaluating the impact of stress ball usage during spinal anesthesia on pain through VAS (Visual Analog Scale) scoresThe VAS score ranges from 0 to 10, with higher values indicating more pain.

SECONDARY OUTCOMES:
Stress ball and blood pressure | Before and after the procedure, at 3 minutes.
  The effect of the stress ball used during spinal anesthesia on the patient's blood pressure.It will be measured before and after the procedure and recorded in mmHg.
Stress ball and pulse | Before and after the procedure, at 3 minutes.
  The impact of the use of the stress ball during spinal anesthesia on the pulse will be assessed.Pulse will be recorded as beats per minute.
Stress ball and saturation | Before and after the procedure, at 3 minutes.
  The impact of using a stress ball during spinal anesthesia on saturation will be evaluated. It will be recorded in percentage.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Özge Sayın Ayan, Istanbul, Eyup
  - Prof.Dr.Cemil Tascioglu City Hospital, Istanbul, Şişli

IPD SHARING:
Plan to Share IPD: Yes
We plan to share the individual participant data (IPD) from this study in two formats: an Excel spreadsheet containing detailed data sets and a PDF document summarizing the key findings. The data sharing is scheduled to occur three months after the completion of the study.
  Data Types and Scope:
  The Excel spreadsheet will encompass comprehensive participant data, covering all relevant variables collected during the study.
  The PDF document will provide a concise summary of the study results, highlighting key outcomes and trends.
Supporting Information: CSR
Time Frame: Approximately 3 months after the completion of the study.
Access Criteria: Access is granted only to individuals with appropriate authorization, such as researchers, healthcare professionals, or authorized personnel.

REFERENCES:
- [Background] Yanes AF, Weil A, Furlan KC, Poon E, Alam M. Effect of Stress Ball Use or Hand-holding on Anxiety During Skin Cancer Excision: A Randomized Clinical Trial. JAMA Dermatol. 2018 Sep 1;154(9):1045-1049. doi: 10.1001/jamadermatol.2018.1783. PMID 30027283
- [Background] Kumar S, Gautam SK, Gupta D, Agarwal A, Dhirraj S, Khuba S. The effect of Valsalva maneuver in attenuating skin puncture pain during spinal anesthesia: a randomized controlled trial. Korean J Anesthesiol. 2016 Feb;69(1):27-31. doi: 10.4097/kjae.2016.69.1.27. Epub 2016 Jan 28. PMID 26885298
- [Result] Hudson BF, Ogden J, Whiteley MS. Randomized controlled trial to compare the effect of simple distraction interventions on pain and anxiety experienced during conscious surgery. Eur J Pain. 2015 Nov;19(10):1447-55. doi: 10.1002/ejp.675. Epub 2015 Jan 30. PMID 25641687